CLINICAL TRIAL: NCT03865771
Title: Sleep Related Memory Consolidation in Children With Age Related Focal Epilepsy.
Acronym: EPIMEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6995
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Benign Epilepsy With Centro Temporal Spikes (BECTS); Atypical Benign Partial Epilepsy (ABPE); Epileptic Encephalopathy With Continuous Spike and Waves During Sleep (ECSWS)
Keywords: Memory consolidation; Epilepsy; Childhood; Benign epilepsy with centro temporal spikes (BECTS); Epileptic encephalopathy with continuous spike and waves during sleep (ECSWS)
MeSH Terms: conditions — Epilepsy | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPILEPSY GROUP (Experimental): Patients with typical BECTS (benign group) or atypical BECTS or ECSWS (severe group)
  Medical visit
  Neuropsychological testing
  Neuropsychological procedure
  Video EEG and polysomnography (standard of care procedure): 2h wake and whole night
  Sleep diary
  Interventions: Behavioral: Neuropsychological testing; Behavioral: Neuropsychological procedure
- CONTROL GROUP (Other): Patients hospitalized for non neurologic illness (diabetes, nephropathy, chronic intestinal disease)
  Medical visit
  Neuropsychological testing
  Neuropsychological procedure
  Video EEG and polysomnography : 2h wake and whole night
  Sleep diary
  Interventions: Behavioral: Neuropsychological testing; Behavioral: Neuropsychological procedure; Other: Video EEG and polysomnography

INTERVENTIONS:
Behavioral: Neuropsychological testing — memory, executive testing, behaviour questionnaire, visual attention,
Behavioral: Neuropsychological procedure — Rey auditory verbal learning test, Delayed recall : 1h, 5h, 24h (after one night sleep)
Other: Video EEG and polysomnography — Video EEG : 10 electrodes + 3 electrodes for PSG 2h wake EEG Whole night EEG
  Arms: CONTROL GROUP

SUMMARY:
Age related focal epilepsies in children encompasses, according to the ILAE criteria, benign epilepsy with centro temporal spikes (BECTS), atypical benign partial epilepsy (ABPE) and epileptic encephalopathy with continuous spike and waves during sleep (ECSWS). These non structural epilepsies are associated with interictal sleep spike and waves activated by sleep. Moreover, high prevalence of learning disorders occur in children with age related epilepsies. A correlation is suspected between learning disorders and sleep activation of spike and waves. The investigators suppose that learning dysfunction is linked to loss of information during sleep of epileptic children, unlike for control patients. As sleep allows memory consolidation of words learned during wakefulness, an epileptic activity during sleep may disrupt this consolidation, leading to a loss of information.

Hypothesis: the investigators hypothesize a disruption of memory consolidation after one night in children affected with ABPE and ECSWS (severe group) compared to memory consolidation in children affected with BECTS (benign group), and control group.

Primary purpose:

To demonstrate that the deficit of delayed recall in 15 word learning test after one night is higher for the "severe group", compared to the "benign group" and the control group.

Secondary purposes:

* to study the evolution over time of memory consolidation
* to evaluate the correlation of the deficit of delayed recall with executive dysfunction, clinical factors of epilepsy, neurophysiological factors of epilepsy, and sleep architecture

ELIGIBILITY:
Inclusion Criteria:

Principal:

* normal psychomotor development
* informed consent signed by both parents and subject if able
* affiliated to social security regimen

Specific

Patients from "severe" and "benign" groups:

* focal age related epilepsy: BECTS, ABPE, ECSWS (ILAE criteria)
* children hospitalized for their follow-up
* normal neuroimaging

Control group

-children hospitalized for a non neurologic disease

Exclusion Criteria:

Principal:

Psychiatric trouble (DSM V) Sensorial trouble without correction Poor command of French language Minor under care

Specific

Patients from "severe" and "benign" groups:

* degenerative disease
* abnormal neuroimaging
* mental deficiency

Control group

* neurologic trouble
* abnormal sleep EEG
* intellectual deficiency

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
memory lapse rate at 24 hours in the severe group, the benign group and the control group. ("memory lapse rate": rate of non recalled words number, during the delayed recall phase of the test, related to the maximal number of words recalled | 24 hours

SECONDARY OUTCOMES:
memory lapse rate for each group | at 1 hour, 5 hours, 24 hours
Correlation of memory lapse rate with Executive functioning tests scores | at 1 hour, 5 hours, 24 hours
Correlation of memory lapse rate with age of onset, epilepsy phase, treatment | at 1 hour, 5 hours, 24 hours
Correlation of memory lapse rate with EEG severity scale, atypical criteria, EEG focus localization, sleep discharges frequency | at 1 hour, 5 hours, 24 hours
Correlation of memory lapse rate with number and organization of sleep cycles | at 1 hour, 5 hours, 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anne DE SAINT MARTIN, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Hopital D'Enfants Pediatrie Medicale Ambulatoire, Nancy
  - Hopital de Hautepierre-Service de Pediatrie/Neurologie, Strasbourg